CLINICAL TRIAL: NCT04609150
Title: Assessment of Vertebral Fat Quantitative MRI as a Marker of Bone Fragility in Patients With Multiple Myeloma
Brief Title: Vertebral Fat Quantitative MRI as a Marker of Bone Fragility in Multiple Myeloma (MYELOMEFRAGIQUANTI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200091
Record Dates: First submitted 2020-10-07; First posted 2020-10-30 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma; Vertebral Fracture
Keywords: Bone marrow fat; Bone fragility; Fat quantification
MeSH Terms: conditions — Multiple Myeloma; Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple myeloma patients with vertebral fractures: Patients followed for multiple myeloma in the Lariboisière/Saint-Louis/Fernand-Widal hospital group, with vertebral fractures treated by vertebroplasty from January 2017 to December 2021, with recent clinical and biological data available at the time of imaging and fracture events
  Interventions: Other: Bone marrow fat quantification by MRI

INTERVENTIONS:
Other: Bone marrow fat quantification by MRI — Bone marrow fat quantification by MRI at the moment of the diagnosis of vertebral fracture before treatment by vertebroplasty

SUMMARY:
Multiple myeloma is a disease that causes increased bone fragility which is often revealed or complicated by vertebral fractures. Invasion of bone marrow by tumor plasma cells leads to bone destruction and reduced fat fraction. The main objective is to assess the correlation between vertebral bone marrow fat fraction and bone fragility represented by a severity score of vertebral fractures. The secondary objective is to assess the correlation with clinical and biological prognostic factors and scores..

DETAILED DESCRIPTION:
Patients treated with vertebroplasty will be included during the period of the study, retrospectively or prospectively.

Mains collected data are represented by :

* Bone marrow fat fraction determined by MRI
* Severity score for vertebral fractures
* Clinical prognostic factors
* Biological prognostic factors
* Clinico-biological scores Descriptive statistics and correlation analyses will be performed between the measured parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed for multiple myelomas in the Lariboisière/Saint-Louis/Fernand-Widal hospital group
* vertebral fractures treated by vertebroplasty from January 2017 to December 2021
* recent clinical and biological data available at the time of imaging and fracture events

Exclusion Criteria:

* Factors modifying the bone marrow fat fraction (extensive radiotherapy)
* Lack of recent clinical or biological data compared to imaging examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for multiple myelomas in the Lariboisière/Saint-Louis/Fernand-Widal hospital group, with vertebral fractures treated by vertebroplasty from January 2017 to December 2021, with recent clinical and biological data available at the time of imaging and fracture events.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of bone marrow fat in vertebral bone marrow | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Measured from Dixon sequences on MRI exams performed in routine care, for the assessment of the relationship between bone marrow vertebral fat content and the severity of the vertebral fractures
Vertebral fracture severity score | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Score established according to morphological criteria determined by MRI/computerized tomography scan, based on the Genant classification. Calculation of sum of the points awarded as follows: vertebral fracture on osteolytic lesion = 3; osteolytic lesion with high fracture risk = 0; other fracture related to increased bone fragility, scale 1-3 according to Genant's criteria, 3 representing the worst situation; normal vertebra = 0.

SECONDARY OUTCOMES:
Sex | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Male or female
Age at the diagnosis of multiple myeloma | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Age in years at the diagnosis of multiple myeloma
Weight/body mass index (BMI) | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  The Body Mass Index is calculated as the ratio between the weight measured in kilograms and the square of the height measured in meters
Age at the moment of the vertebral fracture | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Age in years at the moment of the vertebral fracture
Type of the monoclonal component | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Corresponding the type of the heavy (IgG, IgA, IgD, IgE or IgM) and/or the light chain (κ or λ) of the monoclonal immunoglobulin protein
Serum rate of the monoclonal component | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Serum rate of the monoclonal immunoglobulin protein in g/L
Medullary plasmacytosis | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Percentage of plasma cells assessed by bone marrow aspiration
Presence of anaemia | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Defined by hemoglobin value < 100g/L
Presence of hypercalcemia | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Defined by serum calcium > 2.75mmol/L
Presence of renal failure related to myeloma | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Defined by a creatinine clearance < 40mL/min or serum creatinine > 177µmol/L
Presence of amyloidosis | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Presence of amyloid deposits revealed by tissue biopsy
Multiple myeloma stage according to the Salmon-Durie staging System | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  The Salmon-Durie classification in three stages according to the absence (I) or the presence (III) of the following criteria: anemia (hemoglobin value < 100g/L); hypercalcemia (serum calcium > 2.75mmol/L); amyloidosis (amyloid deposits revealed by biopsy); bone lesion at imaging. Concerning the serum rate of the monoclonal component, IgA < 30g/L and IgG < 50 g/L are considered stage I, and IgA > 50g/L and IgG > 70 g/L are considered stage III. The intermediate stage II is based on the rate of the blood monoclonal component (from 30 to 50 g/L for IgA and from 50 to 70 g/L for IgG) . The subclassification depends on the absence (A) or the presence of renal failure related to myeloma (B) (defined by creatinine clearance < 40mL/min or serum creatinine > 177µmol/L).
Multiple myeloma stage according to the International Staging System (ISS) | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  To determine the International Staging System score (ISS) in three stages with stage I corresponding to serum beta-2-microglobulin < 3.5 mg/L and serum albumin ≥ 35 g/L, stage III corresponding to beta-2-microglobulin ≥ 5.5 mg/L, and stage II when not stage I or III
Serum rate of Lactate dehydrogenase | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Measured in U/L; serum lactate dehydrogenase is a poor prognosis factor when elevated (> 300U/L)
Salmon-Durie Plus classification | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Based of the MRI pattern of multiple myeloma that determine three stages : stage I (0-4 focal lesions), stage II (5-20 focal lesions), stage III (>20 focal lesions). The subclassification depends on the absence (A) or the absence of extramedullary disease (B) (anemia, hypercalcemia, renal failure, amyloidosis)
Type of bone damage on CT scan | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Classified as normal, focal lesion, diffuse osteopenia, focal lesion with diffuse osteopenia
Vertebral radiodensity | At the moment of the diagnosis of the vertebral fracture before treatment by vertebroplasty
  Measured by a CT scan in Hounsfield Units

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BOUSSON, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Lariboisière Hospital, Osteo-Articular, Visceral and Vascular Imaging department, Paris, France

IPD SHARING:
Plan to Share IPD: No